CLINICAL TRIAL: NCT05910190
Title: Effective Use of Buprenorphine for Long-Acting Pain Relief in Combination With Short-Acting Full Agonist Opioids for Cancer Related Pain
Brief Title: Buprenorphine for Cancer Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Principal Investigator, Marcin Chwistek, Director of Supportive Oncology and Palliative Care Program, Fox Chase Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-1060
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Cancer-Related Pain
Keywords: Cancer Pain; buprenorphine
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: prospective, single arm, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Receiving buprenorphine with short acting full agonist opioid with CPM Rx app to document medication use.
  Interventions: Drug: Use of buprenorphine with FAO > 30 OME; Behavioral: CPM Rx application use

INTERVENTIONS:
Drug: Use of buprenorphine with FAO > 30 OME — Patients will receive buprenorphine with concurrent FAO >30 OME and be assessed for withdrawal, pain, and other symptoms.
Behavioral: CPM Rx application use — The CPM Rx application is used on smart phones to allow patients to input time-stamped data about medication type, dosage, and pain score. This will allow analysis of trends in self-reported pain and optimal dosing patterns. Usage over three months will be assessed.

SUMMARY:
This study will evaluate patients on both buprenorphine and full agonist opioids (FAO) to assess for withdrawal symptoms. Patients will be evaluated by clinicians and using validated tools to assess for pain and withdrawal. At the same time, patients will use a CPM Rx application on their phone to track medication use.

DETAILED DESCRIPTION:
This prospective study will recruit patients with pain related to cancer or its treatment who are on buprenorphine in combination with a full agonist opioid where dose of the full agonist opioids (FAO) is > 30 mg OME per day. They will be provided a mobile application (CPM Rx) for reporting of pain level daily and at each as needed dose. Withdrawal will be assessed using a modified Clinical Opioid Withdrawal Scale (COWS) score and patients will be instructed to be aware of changes in these symptoms. They will also be followed in person at the initial visit, and at days 14, 28, 56 , and 84 with Brief Pain Inventory (BPI) and COWS scale to assess for pain or withdrawal and other reported side effects. Pill counts will be done on days 28, 56, and 84 to further assess medication usage. Nurses will check-in to complete BPI and ask about withdrawal symptoms at days 42 and 70. The study seeks to assess if patients on buprenorphine and FAO have withdrawal symptoms, what are the highest doses of buprenorphine and FAO tolerated, and assess usage of the CPM Rx app. Each patient will be followed on the study for 3 months, unless the choose or it is deemed appropriate to end sooner.

ELIGIBILITY:
1. Age greater than or equal to 18 years
2. English speaking and able to understand and sign informed consent and HIPAA consent document.
3. The patient will have pain from any cause with a pain level greater than or equal to 4 on a visual analog scale.
4. The patient will be able to complete study assessments including use of the CPM app (requires Smart Phone)
5. Patients who may become pregnant are using adequate contraceptives.
6. Patient is on the combination of buprenorphine and full agonist opioid > 30 mg oral morphine equivalent or being started on both buprenorphine and full agonist opioid >30 mg oral morphine equivalent at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Withdrawal while on Buprenorphine with Full Agonist Opioids | 3 months
  Patients will be assessed on days 0 (baseline), 14, 28, 42, 56, 70, and 84 to assess for withdrawal using the validated COWS tool in conjunction with clinical assessment.
Maximum dose of FAO with Buprenorphine | 3 months
  Doses of buprenorphine and FAO will be assessed on days 0 (baseline), 14, 28, 42, 56, 70, and 84 with maximum dose of FAO and associated does of buprenorphine and maximum dose of buprenorphine and associated dose of FAO determined at the end of the study.

SECONDARY OUTCOMES:
Usage of CPM Rx | 3 months
  Usage of the app will be monitored and described at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt-Hansen M, Taubert M, Bromham N, Hilgart JS, Arnold S. The effectiveness of buprenorphine for treating cancer pain: an abridged Cochrane review. BMJ Support Palliat Care. 2016 Sep;6(3):292-306. doi: 10.1136/bmjspcare-2015-000939. Epub 2015 Dec 15. PMID 26669324